CLINICAL TRIAL: NCT06438783
Title: A Multicenter, Open-label, Multi-cohort Phase Ib Trial Evaluating the Efficacy and Safety of TQB2928 Injection Combined With Anlotinib Hydrochloride Capsule in Relapsed/Metastatic Osteosarcoma and Other Relapsed/Metastatic Solid Tumors
Brief Title: TQB2928 Injection Combined Anlotinib Hydrochloride Capsule in Recurrent/Metastatic Osteosarcoma and Other Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was closed due to business reasons. Closure was not prompted by any safety or efficacy concerns.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2928-ALTN-Ib-01
Record Dates: First submitted 2024-05-27; First posted 2024-06-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Osteosarcoma; Other Solid Tumors
MeSH Terms: conditions — Osteosarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1200mg of TQB2928 injection +Anlotinib (Experimental): 21 days as a treatment cycle.
  Interventions: Drug: 1200mg of TQB2928 injection+Anlotinib
- 1800mg of TQB2928 injection+Anlotinib (Experimental): 21 days as a treatment cycle.
  Interventions: Drug: 1800mg of TQB2928 injection+Anlotinib

INTERVENTIONS:
Drug: 1200mg of TQB2928 injection+Anlotinib — TQB2928 is a novel humanized immunoglobulin G4 (IgG4) subtype monoclonal antibody targeting Cluster of Differentiation 47 (CD47).
  Arms: 1200mg of TQB2928 injection +Anlotinib
Drug: 1800mg of TQB2928 injection+Anlotinib — TQB2928 is a novel humanized igG4 subtype monoclonal antibody targeting CD47.
  Arms: 1800mg of TQB2928 injection+Anlotinib

SUMMARY:
This is a multicenter, open-label, multi-cohort Phase Ib trial to evaluate the efficacy and safety of TQB2928 injection combined with anlotinib hydrochloride capsule in patients with relapsed/metastatic osteosarcoma and other relapsed/metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of high-grade osteosarcoma(cohort I),dedifferentiated liposarcoma or polytypic liposarcoma(cohort II),unsuitable for local treatment;
* The requirements for front-line treatment received by subjects are as follows:

  1. Subjects with osteosarcoma have failed at least first-line chemotherapy and are not suitable for re-receiving first-line chemotherapy ,or progression within 6 months of the end of first-line therapy;
  2. Subjects with dedifferentiated liposarcoma or polytype liposarcoma who have received at least first-line chemotherapy failure for recurrent/metastatic sites or relapse during postoperative adjuvant chemotherapy or within 6 months after treatment(considered first-line treatment failure).

Exclusion Criteria:

* History of hemolytic anemia from any cause (including Evans syndrome) within 3 months prior to first dosing;
* Subjects with osteosarcoma or dedifferentiated liposarcoma/polytype liposarcoma who have previously used antiangiogenic tyrosine kinase inhibitors (TKI) or bevacizumab or its biosimilar, such as anlotinib, apatinib, lenvatinib, sorafenib, sunitinib, regorafenib, fruquintinib;
* Previous antibody or fusion protein or small molecule drug targeting CD47 or Signal-regulatory protein α (SIRRP-α).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Cohort 1: Progression-Free Survival (PFS) of 6 months | Up to 6 months
  Cohort 1: Kaplan-Meier method was used to plot the survival curve, in which the cumulative survival rate and 95% confidence interval corresponding to the progression-free survival time of 6 months were obtained.
Cohort 2: Overall response rate (ORR) | Up to 6 months
  Cohort 2: The percentage of subjects with complete (CR) or partial response (PR) as determined by the investigator according to the RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Cohort 1: Progression-Free Survival (PFS) of 4 months | Up to 4 months
  Cohort 1: Survival curve was plotted using Kaplan-Meier method. In the curve, the corresponding cumulative survival rate and 95% confidence interval for progression-free survival of 4 months were obtained.
Cohort 1: Overall response rate (ORR) | Baseline up to 96 weeks
  Cohort 1: The percentage of subjects with complete (CR) or partial response (PR) as determined by the investigator according to the RECIST 1.1 criteria.
Cohort 2: Progression-Free Survival (PFS) of 6 months | Up to 6 months
  Cohort 2: Kaplan-Meier method was used to plot the survival curve with the corresponding cumulative survival rate and 95% confidence interval (95% CI) when the progression-free survival time was 6 months. The overall population and 2 dose groups were counted separately (including participants in the safe introduction period and the extended period).
Progression-Free Survival (PFS) of Cohort 1 and Cohort 2 | Up to 96 weeks
  The time between medication or random initiation and objective progression of disease or death from any cause, whichever comes first.
Disease control rate (DCR) of Cohort 1 and Cohort 2 | Up to 6 weeks
  The percentage of subjects with complete response (CR), partial response (PR), or stable disease (SD) for 6 weeks or more as determined by the investigator based on RECIST 1.1.
Duration of response(DOR) of Cohort 1 and Cohort 2 | Baseline up to 96 weeks
  For subjects whose optimal response was complete response (CR) or partial response (PR), defined as from the date when tumor response was first documented to the date when disease progression was first documented or the date of death from any cause, whichever came first.
Overall survival (OS) of Cohort 1 and Cohort 2 | Baseline up to 96 weeks
  From randomization to the time of death from any cause.
Adverse event rate of Cohort 1 and Cohort 2 | Baseline up to 96 weeks
  Incidence and severity of adverse events (AES) and serious adverse events (SAEs), abnormal laboratory test indicators and treatment-related adverse events (TEAEs).
Incidence of Anti-drug antibody (ADA )and Neutralizing Antibody( NAb ) | 30 minutes before administration on day 1 of cycles 1, 2, 4 and 8 (each cycle is 21 days), day 90 after the last administration (±7 days)
  The positive rates of immunogenicity (ADA and NAb) in subjects were summarized and descriptive statistical analysis was performed.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Beijing jishuitan hospital, Beijing, Beijing Municipality
  - Pekjing university people's hospital, Beijing, Beijing Municipality
  - Beijing cancer hospital, Beijing, Beijing Municipality
  - Hunan cancer hospital, Changsha, Hunan
  - Tianjin medical university cancer institute&hospital, Tianjin, Tianjin Municipality